CLINICAL TRIAL: NCT02585726
Title: Lake Washington Vascular VenaSeal™ Post-Market Evaluation: WAVES
Brief Title: Lake Washington Vascular VenaSeal™ Post-Market Evaluation (WAVES)
Acronym: WAVES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lake Washington Vascular (Other)
Collaborators: Syntactx (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-01
Record Dates: First submitted 2015-10-22; First posted 2015-10-23 (Estimated); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Venous Reflux
Keywords: Varicose Veins; Great Saphenous Vein; Venous Insufficiency
MeSH Terms: conditions — Varicose Veins; Venous Insufficiency

ARMS (2):
- Historical Control with Propensity Analysis (Active Comparator)
  Interventions: Device: SP-402 VenaSeal™ Closure System
- VenaSeal Treatment Arm (Experimental)
  Interventions: Device: SP-402 VenaSeal™ Closure System

INTERVENTIONS:
Device: SP-402 VenaSeal™ Closure System — A medical device kit consisting of seven delivery tools and the proprietary VenaSeal™ Adhesive (Medtronic Cardiovascular, Santa Rosa, CA). The device is used to treat venous reflux in lower extremity superficial truncal veins for subjects in the treatment arm..
  Other Names: VenaSeal™

SUMMARY:
The VenaSeal Closure system offers an outpatient treatment option for the permanent closure of lower extremity superficial truncal veins, such as the great saphenous vein (GSV), through endovascular embolization with coaptation. VenaSeal is intended for use in adults with clinically symptomatic venous reflux as diagnosed by duplex ultrasound (DUS).

ELIGIBILITY:
Key Inclusion Criteria:

* Reflux in at least one target vein;
* One or more of the following symptoms related to a TV: aching, throbbing, heaviness, fatigue, pruritus, night cramps, restlessness, generalized pain or discomfort, swelling;
* CEAP classification of C2 (if symptomatic) through C5;

Key Exclusion Criteria:

* Current, regular use of systemic anticoagulation;
* Previous or suspected deep vein thrombosis or pulmonary embolus, or active acute superficial thrombophlebitis, or thrombophlebitis migrans;
* Previous treatment such as laser or radiofrequency ablation of venous disease in targeted vein segment;
* Known hypercoagulable disorder;
* Pregnant or breast feeding at enrollment;
* Known sensitivity to cyanoacrylate adhesives;
* Venous treatment in the contralateral limb within the last 30 days, or who require contralateral treatment within three months;
* Planned to undergo additional ipsilateral treatments on the same leg within 3 months following treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-10; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Complete closure (CC) of the PTVS as assessed by duplex ultrasound 1 month after the index procedure. | 1 month
  CC of the PTVS as assessed by duplex ultrasound 1 month after the index procedure.

SECONDARY OUTCOMES:
CC of the PTVS, as assessed by duplex ultrasound | 1 week and 3 months after treatment
CC of Treated Vein Segments (TVS), expressed on a per-segment basis, as assessed by duplex ultrasound | 1 month and 3 months after the index procedure
Quality of life as measured by the venous clinical severity scores (rVCSS) | 1 and 3 months after treatment
Quality of life as measured by the Aberdeen Varicose Vein Questionnaire (AVVQ) | 1 and 3 months after treatment
Quality of life as measured by the EQ-5D | 1 and 3 months after treatment
Return to normal activities and return to work; day of procedure is day 0 | 1 week, 1 month
Need for adjunctive treatment | 3 months
  Measured in case report form (yes or no, and if yes, the Investigator will specify what the adjunctive measure is).
Safety and adverse event for below the knee greater saphenous vein treatment | 1 week, 1 month, 3 months
Safety and adverse events for large diameter TVS defined as veins larger than 8 mm in diameter | 1 week, 1 month, 3 months
Patient satisfaction | 1 week, 1 month, 3 months
  At selected visits, the subject will complete a brief questionnaire rating satisfaction with treatment provided and whether the subject would undergo the treatment again.
CC of TVS, expressed on a per-segment basis | 1 month and 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Lake Washington Vascular, PLLC, Bellevue, Washington, United States

REFERENCES:
- [Background] Gloviczki P, Comerota AJ, Dalsing MC, Eklof BG, Gillespie DL, Gloviczki ML, Lohr JM, McLafferty RB, Meissner MH, Murad MH, Padberg FT, Pappas PJ, Passman MA, Raffetto JD, Vasquez MA, Wakefield TW; Society for Vascular Surgery; American Venous Forum. The care of patients with varicose veins and associated chronic venous diseases: clinical practice guidelines of the Society for Vascular Surgery and the American Venous Forum. J Vasc Surg. 2011 May;53(5 Suppl):2S-48S. doi: 10.1016/j.jvs.2011.01.079. PMID 21536172
- [Background] Beebe-Dimmer JL, Pfeifer JR, Engle JS, Schottenfeld D. The epidemiology of chronic venous insufficiency and varicose veins. Ann Epidemiol. 2005 Mar;15(3):175-84. doi: 10.1016/j.annepidem.2004.05.015. PMID 15723761
- [Background] van den Bos R, Arends L, Kockaert M, Neumann M, Nijsten T. Endovenous therapies of lower extremity varicosities: a meta-analysis. J Vasc Surg. 2009 Jan;49(1):230-9. doi: 10.1016/j.jvs.2008.06.030. Epub 2008 Aug 9. PMID 18692348
- [Background] Geza M, Gloviczki P. Venous Embryology and Anatomy. In: Bergan JJ, editor. The Vein Book: Elsivier Academic Press; 2007.
- [Background] van Eekeren RR, Boersma D, de Vries JP, Zeebregts CJ, Reijnen MM. Update of endovenous treatment modalities for insufficient saphenous veins--a review of literature. Semin Vasc Surg. 2014 Jun;27(2):118-36. doi: 10.1053/j.semvascsurg.2015.02.002. Epub 2015 Feb 18. PMID 25868763
- [Background] Guex JJ. Endovenous chemical (and physical) treatments for varices: what's new? Phlebology. 2014 May;29(1 suppl):45-48. doi: 10.1177/0268355514526331. Epub 2014 May 19. PMID 24843085
- [Background] Davies HO, Popplewell M, Darvall K, Bate G, Bradbury AW. A review of randomised controlled trials comparing ultrasound-guided foam sclerotherapy with endothermal ablation for the treatment of great saphenous varicose veins. Phlebology. 2016 May;31(4):234-40. doi: 10.1177/0268355515595194. Epub 2015 Jul 9. PMID 26163507
- [Background] El-Sheikha J, Carradice D, Nandhra S, Leung C, Smith GE, Campbell B, Chetter IC. Systematic review of compression following treatment for varicose veins. Br J Surg. 2015 Jun;102(7):719-25. doi: 10.1002/bjs.9788. Epub 2015 Apr 2. PMID 25833417
- [Background] Rasmussen LH, Lawaetz M, Bjoern L, Vennits B, Blemings A, Eklof B. Randomized clinical trial comparing endovenous laser ablation, radiofrequency ablation, foam sclerotherapy and surgical stripping for great saphenous varicose veins. Br J Surg. 2011 Aug;98(8):1079-87. doi: 10.1002/bjs.7555. PMID 21725957
- [Background] Bootun R, Lane TR, Davies AH. The advent of non-thermal, non-tumescent techniques for treatment of varicose veins. Phlebology. 2016 Feb;31(1):5-14. doi: 10.1177/0268355515593186. Epub 2015 Jun 30. PMID 26130051
- [Background] Morrison N, Gibson K, McEnroe S, Goldman M, King T, Weiss R, Cher D, Jones A. Randomized trial comparing cyanoacrylate embolization and radiofrequency ablation for incompetent great saphenous veins (VeClose). J Vasc Surg. 2015 Apr;61(4):985-94. doi: 10.1016/j.jvs.2014.11.071. Epub 2015 Jan 31. PMID 25650040
- [Background] Almeida JI, Javier JJ, Mackay EG, Bautista C, Cher DJ, Proebstle TM. Two-year follow-up of first human use of cyanoacrylate adhesive for treatment of saphenous vein incompetence. Phlebology. 2015 Jul;30(6):397-404. doi: 10.1177/0268355514532455. Epub 2014 Apr 30. PMID 24789750
- [Background] Proebstle TM, Alm J, Dimitri S, Rasmussen L, Whiteley M, Lawson J, Cher D, Davies A. The European multicenter cohort study on cyanoacrylate embolization of refluxing great saphenous veins. J Vasc Surg Venous Lymphat Disord. 2015 Jan;3(1):2-7. doi: 10.1016/j.jvsv.2014.09.001. Epub 2014 Oct 18. PMID 26993674
- [Background] Vasquez MA, Rabe E, McLafferty RB, Shortell CK, Marston WA, Gillespie D, Meissner MH, Rutherford RB; American Venous Forum Ad Hoc Outcomes Working Group. Revision of the venous clinical severity score: venous outcomes consensus statement: special communication of the American Venous Forum Ad Hoc Outcomes Working Group. J Vasc Surg. 2010 Nov;52(5):1387-96. doi: 10.1016/j.jvs.2010.06.161. Epub 2010 Sep 27. PMID 20875713